CLINICAL TRIAL: NCT02348021
Title: BF-14J01 Drug Coated Stent (DCS) Clinical Trial
Brief Title: Leaders Free Japan
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biosensors Europe SA (Industry)
Collaborators: Biosensors Japan Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14J01
Record Dates: First submitted 2014-09-11; First posted 2015-01-28 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease | interventions — Percutaneous Coronary Intervention; Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug Coated Stent (Other): All patients in the one arm will be treated by PCI with the Drug Coated Stent.
  Interventions: Procedure: Percutaneous coronary intervention (PCI); Drug: Dual Anti Platelet Therapy

INTERVENTIONS:
Procedure: Percutaneous coronary intervention (PCI)
Drug: Dual Anti Platelet Therapy — All patients will receive Dual Anti Platelet Therapy for one month

SUMMARY:
Prospective, multi-center, non-randomized, open-label trial designed to enroll 139 patients in Japan. All patients will receive a DCS and will be followed for 2 years.

DETAILED DESCRIPTION:
In this study all patients will receive the a Drug Coated Stent and will receive one month Dual Anti Platelet Therapy.

ELIGIBILITY:
Inclusion Criteria:

Any indication for PCI-S in patients deemed at high risk for bleeding and candidates for 1 month DAPT. This includes candidates with stable angina, silent ischemia, ACS (STEMI and non-STEMI), non-native lesions and in-stent restenosis. Patients must provide written informed consent.

Reasons of unsuitability for > 1 month dual antiplatelet treatment must include one or MORE of the following:

1. Adjunctive oral anticoagulation treatment planned to continue after PCI
2. Age ≥ 75 years old
3. Baseline Hgb <11 g/dl (or anemia requiring transfusion during the 4 weeks prior to enrollment)
4. Any prior intracerebral bleed
5. Any stroke in the last 12 months
6. Hospital admission for bleeding during the prior 12 months
7. Non skin cancer diagnosed or treated < 3 years
8. Planned daily NSAID (other than aspirin) or steroids for >30 days after PCI
9. Planned surgery that would require interruption of DAPT (within next 12 months)
10. Renal failure defined as: Creatinine clearance <40 ml/min
11. Thrombocytopenia (PLT <100,000/mm3)
12. Severe chronic liver disease defined as: patients who have developed any of the following: variceal hemorrhage, ascites, hepatic encephalopathy or jaundice
13. Expected non-compliance to prolonged DAPT for other medical reasons

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Patients expected not to comply with 30 days DAPT
3. Patients requiring a planned staged PCI procedure more than one week after the index procedure
4. Procedure planned to require non-study stents, or stand-alone POBA or stand-alone atherectomy
5. Active bleeding at the time of inclusion
6. Reference vessel diameter <2.25 ~ >4.0mm
7. Cardiogenic shock
8. Compliance with long-term single anti-platelet therapy unlikely
9. A known hypersensitivity or contraindication to aspirin, clopidogrel or other P2Y12 inhibitor (if applicable), stainless steel, zinc, Biolimus A9 or a sensitivity to contrast media, which cannot be adequately pre-medicated
10. PCI during the previous 12 months for a lesion other than the target lesion of the index procedure
11. Participation in another clinical trial (12 months after index procedure)
12. Patients with a life expectancy of < 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Estimated)
Dates: Start 2014-07; Primary Completion 2016-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
The number of patients that experienced either a cardiac death, myocardial infarction and/or a definite/probable stent thrombosis. | 1 year
The number of patients that experienced a clinically driven target lesion revascularization | 1 year

SECONDARY OUTCOMES:
The number of patients that experienced a cardiac death, myocardial infarction and/or a definite/probable stent thrombosis | 2 years
The number of patients that experienced a clinically driven target lesion revascularization | 2 years
The number of patients that experienced a Bleeding per BARC criteria | 30, 60 and 120 days, and 12 and 24 months
The number of patients that experienced a cardiac death | 30, 60 and 120 days, and 12 and 24 months
The number of patients that experienced a definite/probable stent thrombosis. | 30, 60 and 120 days, and 12 and 24 months
The number of patients that experienced a myocardial infarction | 30, 60 and 120 days, and 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — Shonan Kamakura General Hospital
Locations (1):
- Shonan Kamakura General Hospital, Kamakura, Kanagawa, Japan